CLINICAL TRIAL: NCT06710834
Title: Evaluating the Effectiveness of Combining Hemodiafiltration and Hemoadsorption in Comparison to Hemodiafiltration Alone
Brief Title: Comparing Hemodiafiltration with and Without Hemoadsorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Maduell, Head of Dialysis Section, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2024/0704
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Hemodialysis; Hemodiafiltration; Hemoadsorption
Keywords: Adsorption; Convection; Hemodiafiltration; Efficacy
MeSH Terms: interventions — Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemodiafiltration alone (Active Comparator)
  Interventions: Device: Hemodiafiltration
- Hemodiafiltration plus hemoadsorption (Experimental)
  Interventions: Device: Hemoadsorption cartridge; Device: Hemodiafiltration

INTERVENTIONS:
Device: Hemoadsorption cartridge — HA 130 cartridge
  Arms: Hemodiafiltration plus hemoadsorption
Device: Hemodiafiltration — Postdilutional hemodiafiltration

SUMMARY:
Goals: The aim of the study is to assess the efficacy and safety of the combination of HDF + HA compared to HDF. To do this, we will evaluate the elimination of a wide range of molecular weight molecules, including small protein-bound solutes.

Design: Prospective, single-center study. Each patient underwent two dialysis sessions with routine dialysis parameters in which HDF or HDF + HA treatment modality will be compared.

Study subjects: 20 patients, stable on a thrice-weekly hemodialysis program, will be included. Local Ethics Committee will approve the study and patients will give informed consent.

Interventions: Prospective collection of two dialysis sessions. The only difference among the sessions in each patient will be add or no sorbent cartridge. One session with FX60 Cordiax, helixone, Fresenius Medical Care in postdilution on-line hemodiafiltration and another session with the same dialyzer plus HA 130 cartridge. The order of these treatment sessions was randomly. Blood samples for analyses were taken for each patient in the same dialysis session of the week.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (age > 18 years)
* More than 6 months on a dialysis program
* Stable in a hemodialysis program
* AV fistula, prosthesis, or tunneled catheter as vascular access
* No residual diuresis (< 200 ml/day)
* Not enrolled in a living donor transplant program
* No immunosuppressive treatment
* Provide written informed consent

Exclusion Criteria

* Chronic inflammatory diseases
* Neoplasms
* Immunosuppressive treatment or chronic treatment with anti-inflammatory drugs
* Dysfunctional AV fistula or catheter
* Single-needle dialysis
* Kt/V less than 1.3 or PRU < 70%
* Scheduled living donor kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Uremic toxins reduction ratios (RR) | From enrollment to the end of treatment at 4-8 weeks.
  Protein bound uremic toxins: p-cresyl sulfate RR, and indoxyl-sulfate RR. Medium and large molecules: ß2-microglobulin (11,800 Da) RR, myoglobin (17,200 Da) RR, kappa FLC (22,500 Da) RR, prolactin (23,000 Da) RR, α1-microglobulin (33,000 Da) RR, α1-acid glycoprotein (41,000 Da) RR, and lambda FLC (45,000 Da) RR.

SECONDARY OUTCOMES:
Uremic toxins reduction ratios | From enrollment to the end of treatment at 4-8 weeks
  Urea RR (60 Da), creatinine RR (113 Da), and albumin (66,000 Da)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No